CLINICAL TRIAL: NCT02819362
Title: Benefit of a Diagnostic MRI in Case of Pathological Nipple Discharge With Normal Mammography / Ultrasound.
Acronym: IRM-sein
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Société d'Imagerie de la Femme (Other)
Responsible Party: Sponsor
Other Study IDs: IB2013-IRM
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort - MRI: Patients with pathological nipple discharge
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — The magnetic resonance imaging (MRI) will be performed before the two-step surgery: a ductal-MRI sequence (highly weighted sagittal T2) - followed by sequence with axial plane, T2, T1, injection in dynamic sequences, subtractions.

SUMMARY:
Benefit of MRI in pathological nipple discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Single pore nipple discharge neither green nor milky.
2. Mammography (at least 2 shots, +/- centred on retro-areal) normal.
3. Initial ultrasound: normal.
4. Age over 18 years
5. Female
6. Patient affiliated to the social security scheme.
7. Patient information and informed consent signed and dated

Exclusion Criteria:

Physiological milky or green discharge

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathological nipple discharge
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boisserie-Lacroix M, Doutriaux-Dumoulin I, Chopier J, Boyer B, Depetiteville MP, Hoppe S, Brouste V, Chamming's F. Diagnostic accuracy of breast MRI for patients with suspicious nipple discharge and negative mammography and ultrasound: a prospective study. Eur Radiol. 2021 Oct;31(10):7783-7791. doi: 10.1007/s00330-021-07790-4. Epub 2021 Apr 13. PMID 33846843

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Cohort - MRI
Started | 70
Completed | 0
Not Completed | 70
Not completed — On-site MRI could not be performed | 70

BASELINE CHARACTERISTICS:
Population: Population included in the study, satisfying eligibility criteria
Arm/Group | Prospective Cohort - MRI
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 70

OUTCOME MEASURES:

1. Primary Outcome: The Negative Predictive Value (PVV) of MRI
Description: The negative predictive value (NPV) of MRI in patients with pathological nipple discharge with normal mammography / ultrasound.
  The VPN is defined by the ratio: number of patients with a normal histological examination / number of patients with a normal MRI.
Time Frame: At baseline
Population: MRI could not performed as expected (technical problems with the machine - unrelated to the participants or the study). thus MRI data could not be collected, and as such, primary outcome could not be assessed.
Arm/Group | Prospective Cohort - MRI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious and/or Other Adverse Events were not monitored/assessed in this study,
Description: All-Cause Mortality, Serious and/or Other Adverse Events were not monitored/assessed in this study,
Arm/Group | Prospective Cohort - MRI
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes